CLINICAL TRIAL: NCT06350331
Title: Smart Technology Facilitated Patient-centered Venous Thromboembolism Management: A Randomised Controlled Trial
Brief Title: Smart Technology Facilitated Patient-centered Venous Thromboembolism Management
Acronym: SmaVTE-RCT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Navy General Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HZKY-PJ-2024-8-1
Record Dates: First submitted 2024-03-30; First posted 2024-04-05 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Venous Thromboembolism; Digital Health; Health Education
Keywords: Venous Thromboembolism; Mobile Health; Prophylaxis; Health Education
MeSH Terms: conditions — Venous Thromboembolism; Health Education

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mVTEA Management Group (Experimental): Patients randomly assigned to the mVTEA management group will be discharged with mVTEA-assisted patient-centered VTE management.
  Interventions: Other: mobile venous thromboembolism application (mVTEA)
- Routine Management Group (No Intervention): Patients randomly assigned to the routine management group will be given routine post-discharge management in accordance with local clinical practice.

INTERVENTIONS:
Other: mobile venous thromboembolism application (mVTEA) — mVTEA will assist in the management of patients during the post-hospitalization follow-up phase. The mVTEA's doctor terminal automatically sends VTE-related health education materials in different frequencies and contents based on the patient's knowledge of VTE prevention and treatment, as well as their risk of thrombosis and bleeding during follow-up. In addition, thrombosis physicians on the mVTEA's doctor terminal can deliver health education to patients based on their condition. This can be done through the mVTEA doctor-patient communication module, which includes text, photo, and voice interactions.
  Arms: mVTEA Management Group

SUMMARY:
Smart technologies, such as wearable devices, mobile technologies, and artificial intelligence, are being investigated for use in health management. These technologies have the potential to be applied in disease pre-warning, decision-making support, health education, and healthcare maintenance. They are expected to address the challenges in managing thrombosis, improve access to high-quality medical resources in various regions, and enhance the development of a network for thrombosis rescue and treatment prevention.

The objective of this study is to evaluate the impact of mobile venous thromboembolism application (mVTEA) based patient-centered management of venous thromboembolism (VTE) on patients' perceptions of thromboprophylaxis, in order to enhance clinical practice and establish a foundation of evidence for managing patients with VTE.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients ≥18 years of age at admission;
* Previous or current definitive diagnosis of DVT and/or PE by imaging, or at high risk of VTE at discharge: Padua score ≥4 for medical patients and Caprini score ≥5 for surgical patients.
* Signed informed consent

Exclusion Criteria:

* Mental disorder or combination of other serious diseases leading to incapacity for independent living;
* Inability to use smartphones, computer tablets and other smart devices;
* Being pregnant or breastfeeding;
* Have participated in similar trials or are undergoing other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2024-08-17 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
VTE-KAP questionnaire score | The third month after discharge from the hospital
  The VTE-KAP questionnaire is a self-administered questionnaire that includes demographic characteristics, knowledge, attitude, and practice (KAP) of patients towards VTE prevention and treatment. The VTE-KAP questionnaire consists of a total of 53 questions with an overall score range of 41 to 283. The higher the score, the higher the level of knowledge, attitude, and practice. The VTE-KAP questionnaire scores will be evaluated at the third-month follow-up after discharge.

SECONDARY OUTCOMES:
Knowledge, attitude, and practice scores in the VTE-KAP questionnaire | The third month after discharge from the hospital
  The knowledge domain contains 7 questions to assess patients' levels of knowledge regarding VTE prevention and treatment. The total score of knowledge for each study participant ranged from 7 to 53. The attitude domain contains 20 questions to assess patients' attitudes towards VTE prevention and treatment. Each question was scored and the ﬁnal attitude score ranged between 20 and 100. The practice domain contained 26 questions with a score range of 21 to 130 for assessing the implementation of VTE prevention and treatment behaviors in the study patients. The higher the score, the higher the level of knowledge, attitude and practice. The patients' knowledge, attitude, and practice scores in the VTE-KAP questionnaire will be assessed at the third-month follow-up after discharge separately.
Generic quality of life | The third month after discharge from the hospital
  Generic, non-disease-speciﬁc health-related quality of life (QoL) is assessed using the EuroQol 5-Dimension 5-Level (EQ-5D-5L) questionnaire and its corresponding visual analogue scale at the third-month follow-up after discharge. Brieﬂy, the EQ-5D-5L generates an overall index that ranges from 0 (lowest generic QoL) to 1 (highest generic QoL) and is calculated based on country-speciﬁc reference value sets. The EQ-5D-5L health index was calculated with the value set for China. The EuroQol visual analogue scale ranges from 0 to 100, with higher scores indicating better health.
VTE events | 3 months after discharge
  VTE events will be documented during the 3-month follow-up after discharge. VTE events are categorized into three groups: new-onset VTE, hospital-acquired VTE (HA-VTE), and recurrent VTE.
  VTE that occurred for the first time during the study period, including deep vein thrombosis (DVT) and pulmonary embolism (PE), is classified as new-onset VTE.
  HA-VTE is defined as any new-onset VTE that has occurred within 90 days of hospital discharge.
  Recurrent VTE is defined as the appearance of new evidence of VTE after acute VTE has been treated in the acute phase (2 weeks) with significant clinical improvement in signs and symptoms. According to the time of VTE recurrence, it is further categorized into early VTE recurrence (within 3 months after the last VTE occurrence) and late VTE recurrence (more than 3 months after the last VTE occurrence).
Chronic thromboembolic pulmonary hypertension (CTEPH) | The third month after discharge
  The diagnosis of CTEPH will be documented at the third-month follow-up after discharge.
Chronic thromboembolic pulmonary disease (CTEPD) | The third month after discharge
  The diagnosis of CTEPD will be documented at the third-month follow-up after discharge.
Post-pulmonary embolism syndrome (PPES) | The third month after discharge
  The diagnosis of PPES will be documented at the third-month follow-up after discharge.
Major bleeding | 3 months after discharge
  The major bleeding events as defined by the International Society on Thrombosis and Hemostasis (ISTH) will be documented during the 3-month follow-up after discharge.
VTE-related hospitalization | 3 months after discharge
  Hospitalization due to the new-onset DVT and/or PE will be documented during the 3-month follow-up after discharge.
VTE-related rehospitalization | 3 months after discharge
  Rehospitalization due to VTE recurrence, progression, or complications related to VTE treatment will be documented during the 3-month follow-up after discharge.
New-onset of atrial fibrillation or atrial flutter | 3 months after discharge
  The new-onset of atrial fibrillation or atrial flutter will be documented during the 3-month follow-up after discharge.
Death | 3 months after discharge
  Death will be documented during the 3-month follow-up after discharge. It is categorized into all-cause death and PE-related death. All-cause death is defined as death that occurs during the study period, regardless of cause.PE-related death is defined as death that is unequivocally due to PE.

CONTACTS AND LOCATIONS:
Overall Officials: YU-TAO GUO, Doctor, Study Chair — Sixth Medical Center of Chinese PLA General Hospital
Locations (1):
- Sixth Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valerio L, Mavromanoli AC, Barco S, Abele C, Becker D, Bruch L, Ewert R, Faehling M, Fistera D, Gerhardt F, Ghofrani HA, Grgic A, Grunig E, Halank M, Held M, Hobohm L, Hoeper MM, Klok FA, Lankeit M, Leuchte HH, Martin N, Mayer E, Meyer FJ, Neurohr C, Opitz C, Schmidt KH, Seyfarth HJ, Wachter R, Wilkens H, Wild PS, Konstantinides SV, Rosenkranz S; FOCUS Investigators. Chronic thromboembolic pulmonary hypertension and impairment after pulmonary embolism: the FOCUS study. Eur Heart J. 2022 Sep 21;43(36):3387-3398. doi: 10.1093/eurheartj/ehac206. PMID 35484821
- [Background] Klok FA, Ageno W, Ay C, Back M, Barco S, Bertoletti L, Becattini C, Carlsen J, Delcroix M, van Es N, Huisman MV, Jara-Palomares L, Konstantinides S, Lang I, Meyer G, Ni Ainle F, Rosenkranz S, Pruszczyk P. Optimal follow-up after acute pulmonary embolism: a position paper of the European Society of Cardiology Working Group on Pulmonary Circulation and Right Ventricular Function, in collaboration with the European Society of Cardiology Working Group on Atherosclerosis and Vascular Biology, endorsed by the European Respiratory Society. Eur Heart J. 2022 Jan 25;43(3):183-189. doi: 10.1093/eurheartj/ehab816. PMID 34875048
- [Background] Schulman S, Angeras U, Bergqvist D, Eriksson B, Lassen MR, Fisher W; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in surgical patients. J Thromb Haemost. 2010 Jan;8(1):202-4. doi: 10.1111/j.1538-7836.2009.03678.x. Epub 2009 Oct 30. PMID 19878532
- [Derived] Jin ZG, Zhang ZQ, Liu BB, Wang H, Yang Y, Ren LN, Zhang H, Ji W, Zhai ZG, Guo YT. Smart Technology Facilitated Patient-Centered Venous Thromboembolism Management (the SmaVTE Study): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Jun 5;14:e67254. doi: 10.2196/67254. PMID 40473232